CLINICAL TRIAL: NCT07215637
Title: A Multicenter, Open-label, Dose-escalation, Phase Ia/Ib Study to Evaluate the Safety, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of CKD-512 Monotherapy and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Solid Tumor
Brief Title: Phase Ia/Ib Study of CKD-512 Alone and in Combination With Pembrolizumab in Subjects With Advanced or Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: A150_01ST2410
Record Dates: First submitted 2025-09-24; First posted 2025-10-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-10

CONDITIONS: Advanced Solid Tumors; Metastatic Solid Tumors
Keywords: A2aR; adenosine A2A receptor; CKD-512; Advanced Solid Tumors; Metastatic Solid Tumors
MeSH Terms: interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Part A: Monotherapy (Experimental): Dose Level(DL) 1 to DL 6
  Interventions: Drug: CKD-512
- Part B: Combination therapy (Experimental): DL N to DL N+2, combination with Pembrolizumab
  Interventions: Drug: CKD-512; Combination Product: Pembrolizumab

INTERVENTIONS:
Drug: CKD-512 — Orally administered BID
Combination Product: Pembrolizumab — Intravenous (IV) Infusion
  Arms: Part B: Combination therapy

SUMMARY:
The purpose of this first-in-human (FiH) study is to assess the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD), and preliminary efficacy of CKD-512 given alone and in combination with pembrolizumab in subjects with advanced or metastatic solid tumors who have failed all standard available therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed advanced or metastatic solid tumors.
* Progressive disease after or intolerance to standard therapy and no other effective therapeutic options available.
* Measurable disease as defined in Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1).
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Suitable venous access for the study-required blood sampling, including PK and PD sampling.
* Adequate clinical laboratory values and other measures

Exclusion Criteria:

* Active disease involvement of the central nervous system.
* Any serious or life-threatening medical condition unrelated to cancer, psychiatric illness, drug or alcohol abuse, that could, in the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Systemic anticancer treatment within the protocol-specified period prior to the first dose.
* History of any immune-related toxicity that lead to permanent discontinuation of prior anticancer therapy
* Radiation therapy on a limited area is allowed until 4 weeks prior to the first dose of study drug, provided that the radiated lesion is clinically stable.
* Prior treatment with investigational agents ≤21 days before the first dose of study drug(s).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-16 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Part A: Maximum tolerated dose (MTD) or Optimal biologically effective dose (OBED) | Up to 2 years
  Number and proportion of subjects who experience at least 1 DLT based on incidence, nature, and severity of TEAEs and SAEs graded according to NCI-CTCAE version 5.0 as well as on changes from baseline assessments.
Part B: Recommended dose for expansion (RDE) | Up to 2 years
  Number and proportion of subjects who experience at least 1 DLT based on incidence, nature, and severity of TEAEs and SAEs graded according to NCI-CTCAE version 5.0 as well as on changes from baseline assessments.

SECONDARY OUTCOMES:
Safety and tolerability | Up to 2 years
  Incidence and severity of TEAEs, incidence of SAEs and TRAEs etc. according to the NCI-CTCAE version 5.0
Maximum Observed Plasma Concentration (Cmax) | Up to 2 years
  Cmax is defined as the maximum observed plasma concentration of CKD-512
Cmax at steady state (Cmax_ss) | Up to 2 years
  Cmax_ss is defined as the maximum observed plasma concentration of CKD-512 at steady state
Area Under the Curve to the last measurable concentration (AUClast) | Up to 2 years
  AUClast is defined as the area under the plasma concentration-time curve of CKD-512 from the time of dosing to the time of the last measurable concentration.
Area Under the Curve over the dosing interval tau (AUCtau) | Up to 2 years
  AUCtau is defined as the area under the plasma concentration-time curve of CKD-512 over a dosing interval (tau), usually at steady state.
Overall Response Rate (ORR) | Up to 2 years
  ORR is defined as the percentage of participants whose best overall response is either complete response (CR) or partial response (PR), assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
Duration of Response (DOR) | Up to 2 years
  DOR is defined as the time from the date of the first documented objective tumor response (CR or PR) assessed according to RECIST or iRECIST criteria, until the date of the first documented disease progression or death from any cause, whichever occurs first.
Disease Control Rate (DCR) | Up to 2 years
  DCR is defined as the percentage of participants whose best overall response is CR, PR, or stable disease (SD), assessed according to RECIST version 1.1 or iRECIST criteria.
Progression-Free Survival (PFS) | Up to 2 years
  PFS is defined as the time from the date of treatment initiation to the date of the first documented disease progression or death from any cause, whichever occurs first, assessed according to RECIST version 1.1 or iRECIST criteria.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Yonsei University Health System, Seoul, South Korea